

## **Clinical Development**

#### KJX839/Inclisiran

#### CKJX839A1GB01 / NCT04807400

A phase IIIb, multicentre, randomised controlled study to evaluate the implementation, preference and utility for administration of inclisiran sodium in participants with Atherosclerotic Cardiovascular Disease (ASCVD) or ASCVD-risk equivalents and elevated Low Density Lipoprotein Cholesterol (LDL-C) using a primary care models in the NHS

# **Statistical Analysis Plan (SAP)**

Author:

Document type: SAP Documentation

Document status: Amendment v1.1

Release date: 15-May-2023

Number of pages: 37

Property of Novartis
Confidential
May not be used, divulged, published or otherwise disclosed without the consent of Novartis

Template Version 4.0, Effective from 23-Apr-2021

# **Document History – Changes compared to previous final version of SAP**

| Date | Time point | Reason for update | Outcome for update | Section and title impacted (Current) |
|---|---|---|---|---|
| 31-Mar-<br>2023 | Prior to DB lock | Creation of final version 1.0 | N/A – First version | NA |
| 15-May-<br>2023 | Prior to DB lock | Creation of amendment 1 version 1.1 | <ul> <li>Updated number of imputations from 100 to 500</li> <li>Removed text related to line plot</li> <li>Added clarification text about baseline imputation values in sensitivity analysis</li> </ul> | Section 2.5.2<br>Section 5.5.1 & 5.5.2<br>Section 2.5.5 |
| | | | • Added clarification text | Section 2.10.1<br>Section 5.4 |
| | | | • Other minor format changes | Section 2.5.2 & 2.6.2 |

#### **Table of contents** 1.1 1.2 Study objectives, endpoints and estimands ......9 2.1 2.1.1 2.2 2.2.1 2.3 2.3.1 2.3.2 2.3.3 2.4 Treatments (study treatment, rescue medication, concomitant therapies, 2.4.1 2.4.2 2.5 Analysis supporting primary objective(s)......15 2.5.1 2.5.2 2.5.3 2.5.4 2.5.5 2.5.6 2.6 2.6.1 2.6.2 Statistical hypothesis, model, and method of analysis......21 2.6.3 2.7 2.7.1 2.7.2 Deaths......24 2.7.3 Laboratory data ......24 2.7.4 Other safety data ......24 2.8

| | | 2.8.1 | The CSQ-8 PROMs Questionnaire | 24 |
|---|---|---|---|---|
| | | 2.8.2 | The PAM PROMs Questionnaire | 24 |
| | | 2.8.3 | | |
| | 2.9 | | | |
| | 2.10 | | | |
| | 2.11 | Interim | analysis | 26 |
| 3 | Samp | le size ca | lculation | 26 |
| 4 | Chang | ge to prot | tocol specified analyses | 26 |
| 5 | | | | |
| | 5.1 | Imputa | tion rules | 26 |
| | | 5.1.1 | Study drug | 26 |
| | | 5.1.2 | AE date imputation | 27 |
| | | 5.1.3 | Concomitant medication date imputation | 28 |
| | 5.2 | AEs co | ding/grading | |
| | 5.3 | | criteria for AE of special interest | |
| | 5.4 | Labora | tory parameters derivations | 30 |
| | 5.5 | Statisti | cal models | 31 |
| | | 5.5.1 | Multiple Imputation Wash-out model | 31 |
| | | 5.5.2 | Imputation of undetectable data | 33 |
| | 5.6 | Rule of | f exclusion criteria of analysis sets | 34 |
| 6 | Refer | ence | | 36 |
| | st of t | ables | A malurain review decrees from a rate and a deal and review t | 12 |
| | ble 2-1 | | Analysis windows for each scheduled visit | |
| | ble 5-1 | | Clinical notable criteria for selected laboratory tests | |
| | ble 5-2 | | Notable Liver function test values | |
| | ble 5-3<br>ble 5-4 | | Range determination | |
| Iа | nie $3-4$ | | Projecti deviation criteria leading to exclusion from analysis sets | 44 |

## List of abbreviations

| List of apprevi | |
|---|---|
| AE(s) | Adverse event(s) |
| ALP | Alkaline phosphatase |
| ALT | Alanine aminotransferase |
| AST | Aspartate aminotransferase |
| ASCVD | Atherosclerotic Cardiovascular Disease |
| ATC | Anatomical Therapeutic Chemical |
| CFIR | Consolidated Framework for Implementation Research |
| CRO | Contract Research Organization |
| CSQ-8 | Client Satisfaction Questionnaire |
| CSR | Clinical Study Report |
| CTC | Common Terminology Criteria |
| DBL | Direct Bilirubin |
| ECG | Electrocardiogram |
| EMR | Electonic Medical Record |
| EOS | End of Study |
| - 1 cm | European Union Drug Regulating Authorities Clinical Trials |
| EudraCT | Database |
| eGFR | Estimated glomerular filtration rate |
| EudraCT | European Union Drug Regulating Authorities Clinical Trials |
| FAS | Full Analysis Set |
| HbA1C | Hemoglobin A1c |
| HDL-C | High density lipoprotein cholesterol |
| LDL | Low density lipoprotein |
| LDL-C | Low density lipoprotein cholesterol |
| MAR | Missing at random |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MMRM | Mixed-effect model for repeated measures |
| MNAR | Missing not at random |
| NICE | National Institute for Health and Care Excellence |
| PAM | Patient Activation Measure |
| PT | Preferred term |
| PROM | Patient Reported Outcome Measure |
| RAN | Randomized set |
| REML | Restricted Maximum Likelihood |
| | Testivos itaminismi Emerimova |
| S.C. | Subcutaneous |
| SAE | Serious adverse event |
| SAF | Safety analysis set |
| SAP | Statistical Analysis Plan |
| ~111 | - amionom i manjono i min |

| SCR | Screened set |
|---|---|
| SD | Standard deviation |
| SMC | Scottish Medicines Consortium |
| SMQ | Standardized MeDRA Query |
| SOC | System Organ Class |
| SPIRIT | Study in Primary care evaluating Inclisiran deliveRy Implementation + enhanced SupporT |
| TBL | Total Bilirubin |
| TEAE | Treatment emergent adverse event |
| ULN | Upper limit of normal |

#### 1 Introduction

This document includes the analysis details of study CKJX839A1GB01. Data will be analyzed according to section 12 (data analysis and statistical methods) of CKJX839A1GB01 amended protocol v02 dated 12-Sep-2022.

The efficacy and safety analyses will be conducted after all participants have completed the Day 270 visit or discontinued prior to the Day 270 visit. There is no interim analysis planned for this study. The final analyses will be conducted when the trial has ended, and the results will be summarized in the final CSR.

The analysis of Process Evaluation Sub-study data is out of scope of this SAP.

#### 1.1 Study design

A phase IIIb, multicentre, randomised controlled study to evaluate the implementation, preference and utility for administration of inclisiran sodium in participants on established lipid lowering medication or, have been recommended lipid lowering therapy by their healthcare provider but are unable to tolerate treatment, with elevated low density lipoprotein cholesterol (LDL-C) in a primary care population.

This study is an implementation research study that utilises implementation science methodology with the primary focus being implementation and 'transactability' – how to organise, deliver and maintain an innovative treatment for ASCVD in a primary care setting in a sustainable way.

900 eligible participants will be randomised (300 per treatment group) at up to 30 primary care centres across Greater Manchester.

At the baseline visit/screening on receipt of a signed consent form, eligible participants will be randomised to one of the three treatment groups:

- **Group 1:** Participants will continue to receive their background lipid lowering therapy plus behavioural support
- **Group 2:** Participants will continue to receive their background lipid lowering therapy, plus inclisiran for injection (delivered in an injection-only model).
- **Group 3:** Participants will continue to receive their background lipid lowering therapy, plus inclisiran for injection, plus behavioural support.

Subjects in treatment group 1 will be referred to as the control group in this study.

The study duration will be approximately 9 months. There are no interim analyses planned for this study.

#### Schematic of study design



For elaborated details on study design please refer to the study design section of the protocol.

#### Study objectives, endpoints and estimands 1.2

| Objective(s) | Endpoint(s) |
|---|---|
| Primary objective(s) | Endpoint(s) for primary objective(s) |
| • The primary objective of this study is to demonstrate superiority of inclisiran +/- behavioural support compared to standard of care + behavioural support in a primary care setting, in terms of the percentage change in LDL-C from baseline to Day 270 in adults with elevated LDL-C. | Percentage change in LDL-C from baseline to Day 270. |
| Secondary objective(s) | Endpoint(s) for secondary objective(s) |
| The secondary objectives of this study are to evaluate the implementation of inclisiran +/-behavioural support compared to standard of care + behavioural support in a primary care setting using the following assessments: | |
| Measures of patient satisfaction using the<br>validated CSQ-8 (Client Satisfaction<br>Questionnaire) administered after<br>treatment at day 90. | • Mean difference in total score using the validated CSQ-8 (Client Satisfaction Questionnaire) administered after treatment at day 90. |
| Measures of patient activation and<br>empowerment using the validated Patient<br>Activation Measure (PAM) questionnaire<br>administered after treatment at day 90. | Mean difference in total score using the validated Patient Activation Measure (PAM) questionnaire administered after treatment at day 90. |
| Measures of adherence to cardiovascular disease self-management using the validated Patient Activation Measure (PAM) questionnaire administered after treatment at day 90 and using assessment of medication adherence during the study period. | • The frequency and percentages of subjects in the four levels of the PAM scores (below) will be summarized. Highly activated patients (level 3 and level 4) are more likely to adhere to cardiovascular self-management and thus medication adherence. |
| | Level 1: Disengaged and overwhelmed |
| | Level 2: Become aware but still struggling |
| | Level 3: Taking action |

| | Level 4: Maintaining behaviors and pushinng further. |
|---|---|
| <ul> <li>A process evaluation conducted using the Consolidated Framework for Implementation Research (CFIR) which will explore inclisiran delivery at three levels:</li> <li>Level 1: Feasibility and acceptability of delivery models for inclisiran to patients</li> <li>Level 2: Feasibility and acceptability of</li> </ul> | This SAP does not intend to describe methodology adopted for the Process Evaluation Sub-study data analysis. This study objective is listed for completeness only. For further detail on the process evaluation and planned analyses, please refer to section 4.3 of the Protocol. The analysis results will be reported in final CSR. |
| delivery models for inclisiran to providers (inner setting) | |
| 3. <b>Level 3:</b> Wider 'transactability' of the proposed delivery models (outer setting) | |
| 4. The service costs of each delivery model | |
| 5. The acceptability and perceived sustainability of patient identification and referral routes | |
| Data from the process evaluation will initially analysed blind to trial outcomes (this analysis will then be used to compare and explain any differences in outcomes between intervention arms). | |
| Serious adverse event profile | • Incidence, severity and relationship to<br>the study drug of treatment emergent<br>adverse events, serious adverse events<br>and adverse events leading to treatment<br>discontinuation. |
| | • Incidence of on-treatment and post-treatment deaths. |



#### 2 Statistical methods

#### 2.1 Data analysis general information

All analyses will be performed by Novartis or a designated CRO. The most recent version of SAS available in the statistical programming environment of Novartis or the designated CRO will be used for the analysis.

Final analysis will be conducted after all participants either complete the study or discontinued early. Final analyses will be reported in Final CSR.

Additional analysis may be conducted to evaluate the impact of COVID-19 pandemic, if required.

#### 2.1.1 General definitions

#### Study day:

Study day will be defined as the number of days since the date of first dose of study treatment. The date of first dose of study treatment will be defined as Day 1 and the day before the first dose of study treatment will be defined as Day -1.

Therefore, for a particular date, study day will be calculated as follows:

For dates on or after the first date of study treatment,

Study day = Assessment date - Date of first dose of study treatment + 1;

For dates prior to the first date of study treatment,

Study day = Assessment date – Date of first dose of study treatment.

In case, participant has been randomized but has not received study treatment then randomization visit day will be considered as Day 1.

#### **Baseline definition:**

The baseline assessment is defined as the last non-missing assessment (scheduled or unscheduled) collected before the first dose of study treatment (Day 1) or randomization visit day, if no study treatment has been received.

#### **Post-baseline measurement:**

Post-baseline values are defined as those measurements that were collected after the first dose of study treatment or randomization visit if no study treatment has been received.

When change from baseline is of interest the following formula will be used for each scheduled visit and time-point where baseline and post-baseline values are both available:

Change from baseline = post-baseline value – baseline value.

Percent change from baseline = (change from baseline / baseline value)\*100.

#### **Visit windows:**

If there is more than one observation in a specific window, then the one closest to the target day will be used for analysis. If there are two or more observations that are equally distant to the target day and within the analysis window, the first of these observations will be selected for analysis. Observations that are out of the analysis window below will be classified as unscheduled visits and will not be included in the primary and key secondary efficacy analysis. However, all data will be included in the subject data listings.

As shown in the table below, all visit will apply a window of  $\pm$  14 days.

Table 2-1 Analysis windows for each scheduled visit

| Visit Name | Target day | Analysis window |
|--------------------|------------|-----------------|
| Screening/Baseline | -1 | Day -14 to -1 |
| Visit 1 | 1 | Day 1 to 14 |
| Visit 2 | 90 | Day 76 to 104 |
| End of Study | 270 | Day 256 to 284 |

<sup>\*</sup>Day 1 is defined as day of initiation of study drug administration or randomization visit day if no study treatment has been received.

#### 2.2 Analysis sets

Screened Set (SCR) will include all participants who provided study informed consent.

Randomized set (RAN) will consist of all participants who received a randomization number, regardless of whether study treatment received or not.

Full Analysis Set (FAS) will consist of all randomised participants with the exception of those mis-randomised participants who did not receive study drug. Mis-randomised participants are defined as not qualified for randomisation and are inadvertently randomised into the study. According to the intent to treat principle, participants will be analysed according to the treatment they have been assigned to during the randomisation procedure. The FAS will be used in analyses for the primary, secondary,

**Safety Set (SAF)** will consist of all participants who received at least one dose of study treatment. Participants will be analysed according to the study treatment received. This will be the primary population for the safety analyses.

#### 2.2.1 Subgroup of interest

No subgroup analysis is planned.

# 2.3 Patient disposition, demographics and other baseline characteristics

#### 2.3.1 Patient disposition

The overall number of participants who entered, completed, and discontinued the study will be summarized and listed, including the reasons for discontinuation. Duration on study is defined as: date of last known visit on study – date of first dose of treatment/randomization visit, if no study treatment has been received.

The duration on study will be summarized by treatment group. The screening disposition will be based on SCR. The FAS will be used for the summary and listing of patient disposition. The number of participants in the FAS will be summarized by treatment group. Number of participants with protocol deviations will be tabulated by category (e.g., selection criteria not met, subject not withdrawn as per protocol, treatment deviation, prohibited concomitant medication, other), deviation using FAS. Listing of participants with protocol deviation will be provided.

The number of participants included in each analysis set will be tabulated using RAN. Participants exclusion from analysis sets will be summarized for all patients with reasons for exclusion (i.e. including both protocol and non-protocol deviations) and corresponding listing will be provided.

#### 2.3.2 Demographics and other baseline characteristics

| Demographic and other basel | line data including age, race, | , gender, baseline characteristics such |
|---|---|---|
| as body height, | smoking history, Dietary a | dvice status, Exercise status; baseline |
| disease characteristics like I | DL-C, baseline use of other | er lipid-lowering therapies (yes, no), |
| statin intolerance history(yes, | , no), baseline diabetes status | s determined by the fasting glucose (> |
| 7.0 mmol/L) or random glue | $cose (\geq 11.1 mmol/L) or H$ | bA1C ( $\geq 6.5\%$ or 48 mmol/mol) or |
| medical history, baseline mea | asurements | will be summarized descriptively by |
| treatment group for FAS. Lis | tings will also be provided. | |

Categorical data will be presented as frequencies and percentages by treatment group. For continuous data, non-missing observations, mean, standard deviation, median, 1st and 3rd quartile, minimum, and maximum will be presented.

No inferential statistics will be provided for baseline comparability among the treatment groups.

In addition, the following categorizations of continuous variables will be done:

- Age groups  $< 65, \ge 65 \text{ and } < 75, \ge 75$
- LDL-C subcategories Category 1:  $\leq$  2.6 mmol/L, > 2.6 mmol/L; Category 2:  $\leq$  2.1 mmol/L, > 2.1  $\leq$  2.6 mmol/L, > 2.6  $\leq$  3.3 mmol/L and > 3.3 mmol/L
- •

#### 2.3.3 Medical History

Relevant medical histories and current medical conditions at baseline will be summarised separately by system organ class and preferred term, by treatment group. Histories of statin intolerance will be summarised by treatment group. FAS will be used for the analysis.

# 2.4 Treatments (study treatment, rescue medication, concomitant therapies, compliance)

All summaries of treatments will be performed on the Safety Set, unless otherwise specified.

#### 2.4.1 Study treatment / compliance

The number of study doses administered, duration of exposure, patient year of exposure will be summarized by treatment group. Listings will be provided.

The number of participants dosed will also be summarized by study visit and treatment group.

Duration of exposure for inclisiran arms will be calculated as: minimum of (Date of last dose of treatment – Date of first dose of treatment + 180, Date of last known visit – Date of first dose of treatment).

Duration of exposure for lipid lowering therapies will be calculated as: minimum of (Date of last dose of lipid lowering therapy – Date of first dose of lipid lowering therapy, Date of last known visit – Date of first dose of lipid lowering therapy).

Patient-year of exposure will be calculated as duration of exposure/365.25.

#### 2.4.2 Prior, concomitant and post therapies

Medications are collected through EMR and in this system medication end date is not available.

Lipid-lowering therapy use at screening and baseline/randomization visit (Day 1) will be summarized by treatment group. Lipid-lowering therapy newly added or changed after randomization will be summarized by treatment group.

Other medications will be listed and summarized according to the anatomical therapeutic chemical (ATC) classification system and preferred term, by treatment group.

#### 2.5 Analysis supporting primary objective(s)

The primary objective of this study is to demonstrate superiority of inclisiran +/- behavioural support compared to standard of care + behavioural support in a primary care setting, in adults with elevated LDL-C. Standard of care + behavioural support will be considered as control group as mentioned in section 1.1.

#### 2.5.1 Primary endpoint(s)

The primary endpoint is the percentage change in LDL-C from baseline to Day 270.

The primary estimand is defined as follows. The primary effectiveness question of interest is: What is the effect of the test treatment inclisiran versus control on change in LDL-C after 270 days of treatment in adults on established lipid lowering medication or who have been recommended lipid lowering therapy by their health care provider but are unable to tolerate treatment, regardless of treatment discontinuation for any reason and regardless of unforeseen change in the concomitant lipid lowering therapy.

The justification for the primary estimand is that it will capture both the effect of the study drug and the effect of changes in additional medication(s) used for lipid lowering, if they occur, in a primary care setting.

The primary estimand is described by the following attributes:

| Population | Adults with elevated LDL-C on established lipid lowering medication or, have been recommended lipid lowering therapy by their health care provider but are unable to tolerate treatment. |
|---|---|
| Variable | Percentage change in LDL-C from baseline to Day 270 |
| Treatment | The randomised treatment (inclisiran alone or inclisiran with behavioural support) as add-on to the control treatment of lipid-lowering background therapy plus behavioural support, regardless of treatment discontinuation for any reason and regardless of unforeseen change in the concomitant lipid lowering therapy and regardless of use of prohibited medications. |
| Summary measure | Difference between treatments in mean percentage change in LDL-C from baseline to Day 270. |
| Intercurrent events | <ol> <li>Study treatment discontinuation</li> <li>Deviation in background treatment</li> <li>Use of prohibited medications</li> </ol> |

Patients who took extra dose of inclisiran (who are identified through EMR) during the study period will be excluded and additional analysis will be provided.

#### 2.5.2 Statistical hypothesis, model, and method of analysis

The primary effectiveness objective of this study is to demonstrate superiority of each inclisiran arm compared to control in terms of the percentage change from baseline in LDL-C to Day 270 in adults with elevated LDL-C. The statistical hypotheses that will be tested for each inclisiran arm are as follows:

- H<sub>0</sub>: The difference between participants treated with inclisiran and control in the least squares mean percentage change from baseline to the Day 270 visit in LDL-C= 0
- H<sub>a</sub>: The difference between participants treated with inclisiran and control in the least squares mean percentage change from baseline to the Day 270 visit in LDL-C < 0

The primary objective will be achieved if null hypothesis (H<sub>0</sub>) rejected at the one-sided significance level of 0.025.

The primary analysis will use an analysis of covariance (ANCOVA) model on the percent change in LDL-C from baseline to Day 270 to test the superiority of inclisiran over control after missing data imputation.

Due to probable heterogeneity of variances between treatment groups, ANCOVA model which assumes unequal variances for treatment group will be used. The model will include the fixed effects of treatment group with baseline LDL-C as a covariate.

Multiple imputation will be used to impute missing data using a washout model specified in Appendix 5.5.1. A total of 500 imputed datasets will be created. The ANCOVA model will be fitted to each imputed dataset, and results will be combined using Rubin's combination rules. The estimate and corresponding 2-sided 95% confidence intervals of mean difference between treatment groups will be calculated. p-value for hypothesis test for mean difference will also be provided. The FAS will be used for this analysis. The family-wise error rate for comparisons of the two inclisiran arms with the lipid-lowering background therapy plus behavioural support arm will be controlled using the Holm procedure.

#### 2.5.3 Handling of intercurrent events

The approach of accounting for intercurrent events is as follows:

Primary estimand:

| Intercurrent events (ICEs) | Strategy and justification of handling ICEs | Missing value imputation |
|---|---|---|
| Study<br>treatment<br>discontinuation | Here interest is in effect of treatment regardless of treatment discontinuations due to any reasons other than intercurrent event. This event will be handled using a treatment policy strategy. | The LDL-C data collected post discontinuation of study treatment will be included in the analysis. If there is no off-treatment data available, then missing data on Day 270 or after treatment discontinuation will be imputed using missing not at random (MNAR) for inclisiran arms and using missing at random (MAR) |

| Intercurrent events (ICEs) | Strategy and justification of handling ICEs | Missing value imputation |
|---|---|---|
| | | approach for placebo arm participants. |
| Deviation in background treatment | Interest is in effect of treatment regardless of substantial changes to background therapy during study treatment. This will be handled with a <b>treatment policy strategy</b> . | The LDL-C data collected after deviation in background treatment will be included in the analysis. Missing values will be imputed in same way as mentioned in Appendix 5.5.1 |
| Use of prohibited medications | Interest is in effect of treatment regardless of changes in concomitant lipid lowering medication during study treatment. This will be handled with a treatment policy strategy. | The LDL-C data collected after deviation in background treatment will be included in the analysis. Missing values will be imputed in same way as mentioned in Appendix 5.5.1 |

#### 2.5.4 Handling of missing values not related to intercurrent event

The point of care device is used to measure lipid profile data at each visit. Any undetectable calculated LDL-C data due to device sensitivity for a lipid parameter will be considered as missing for the primary analysis.

Undetectable data will be imputed separately as per Appendix 5.5.1 and used in a sensitivity analysis.

LDL-C data will be calculated using Friedwald's formula as mentioned below:

LDL-C = Total cholesterol – HDL – Triglycerides/2.2

Friedewald's formula valid only when Triglycerides < 4.52 mmol/L



Other missing data are expected to be intermittent missing data and will be assumed to be missing at random. The post-death missing values will be treated in same way as other missing data. Imputation details for data missing at random in the washout model has been provided in Appendix 5.5.1.

#### 2.5.5 Sensitivity analyses

The following sensitivity analyses will be performed for the primary estimand, to assess the robustness of the estimation in the presence of deviations from the assumptions specified in the primary analysis on the FAS only:

• Linear mixed-effect model for repeated measures (MMRM) analysis without multiple imputation

Analyses using the MMRM will include fixed effects for treatment, visits, interaction between treatment and visits, baseline LDL-C and interaction between baseline LDL-C and visit. Day 90 and 270 will be included as visit. The Restricted Maximum Likelihood (REML) estimation approach will be used with covariance structure set as "Unstructured". If the model does not converge with unstructured covariance matrix, the compound symmetry covariance matrix will be used in the mixed model.

As a sensitivity analysis, the imputation algorithm will be changed from a regression approach to a multivariate normal model to include in the imputation information that is provided by undetectable LDL-C values. An LDL-C value is undetectable when either are outside of the limit of detection. Based on the limit of detection and through Friedewald's formula, a range for an LDL-C value can be calculated. In this sensitivity analysis, the LDL-C range is considered in the imputation model. As for the primary analysis, undetectable LDL-C values for either study arm are imputed under a MAR assumption, missing values in the placebo arm are imputed under a MAR assumption, and missing data on Day 270 or after treatment discontinuation in the inclisiran arm are imputed using a wash-out model (i.e., using a jump-to-reference approach).

In the sensitivity analysis, imputed baseline values will be restricted to  $\geq 0.1$  to avoid imputed values close to zero which can lead to numerical instabilities in the analysis of percentage LDL-C change from baseline.

The imputation will be carriedout using in SAS/R as mentioned in Appendix 5.5.2.

The analysis will be carried out using ANCOVA procedure as mentioned in section 2.5.2.

#### 2.5.6 Supplementary analyses

Supplementary analysis of LDL-C change from baseline to Day 270 will be performed using linear mixed-effect model for repeated measures (MMRM) analysis with multiple imputation as specified in section 2.5.5. This supplementary analysis will be performed by assessing supplementary estimand as mentioned below.

Intercurrent events (Study treatment discontinuation and Deviation in background treatment) will be handled similarly as mentioned in primary endpoint (Refer section 2.5.3) and additionally below mentioned strategy will be used for "Use of prohibited medications".

| ICE | Strategy and justification of handling ICEs | Missing value imputation |
|---|---|---|
| Use of prohibited medications | Interest is in effect of treatment regardless of changes in concomitant lipid lowering medication during study treatment. Use of prohibited medications (includes treatments which are | LDL-C data after this event will be set to missing. Missing data after this event will be imputed in same way as mentioned in Appendix 5.5.1. |

| ICE | Strategy and justification of handling ICEs | Missing value imputation |
|---|---|---|
| | added to existing background therapy during the study) will not be allowed in the study and will lead to study treatment discontinuation. | |
| | The LDL-C data collected after the use of any prohibited medication will not be included in the analysis. | |
| | Hypothetical strategy with the hypothetical scenario 'as if patients would have not received any prohibited medication. | |

#### 2.6 Analysis supporting secondary objectives

The secondary objectives of this study are to evaluate the implementation of inclisiran +/-behavioural support compared to standard of care + behavioural support in a primary care setting using the following assessments that will be reported based on this SAP are:

- Measures of patient satisfaction using the validated CSQ-8 (Client Satisfaction Questionnaire) administered after treatment at day 90.
- Measures of patient activation and empowerment using the validated Patient Activation Measure (PAM) questionnaire administered after treatment at day 90.
- Measures of adherence to cardiovascular disease self-management using the validated Patient Activation Measure (PAM) questionnaire administered after treatment at day 90 and using assessment of medication adherence during the study period.
- Serious adverse event profile and adverse events leading to treatment discontinuation.

The following secondary endpoint will be analysed by Manchester University and are not covered by this SAP:

- A process evaluation conducted using the Consolidated Framework for Implementation Research (CFIR) which will explore inclisiran delivery at three levels:
  - Feasibility and acceptability of delivery models for inclisiran to patients
  - > Feasibility and acceptability of delivery models for inclisiran to providers (inner setting)
  - Wider 'transactability' of the proposed delivery models (outer setting)
  - ➤ The service costs of each delivery model
  - > The acceptability and perceived sustainability of patient identification and referral routes

#### 2.6.1 Secondary endpoint(s)

The following are key secondary efficacy endpoints:

- Mean difference in total score using the validated CSQ-8 (Client Satisfaction Ouestionnaire) administered after treatment at day 90.
- Mean difference in total score using the validated Patient Activation Measure (PAM) questionnaire administered after treatment at day 90.
- Measures of adherence to cardiovascular disease self-management using the validated Patient Activation Measure (PAM) questionnaire administered after treatment at day 90 and using assessment of medication adherence during the study period.

All the analyses on above endpoints will be based on observed data only.

#### 2.6.1.1 The CSQ-8 PROMs Questionnaire

The Client Satisfaction Questionnaire<sup>©</sup> (CSQ) is a portfolio of measurement instruments (CSQScales<sup>®</sup>) designed to assess consumer satisfaction with health and human services, including governmental and public benefit programs and services.

Each scale measures the recipients' direct satisfaction with specific services offered and received within a particular time frame from a specific provider or service setting.

The CSQ-8 has 8 items and no subscales. and It reports a single score measuring a single dimension of overall satisfaction.

A total score is produced by summing all item responses, with a higher scores indicating higher satisfaction. The outcome is the mean difference in total score between treatment groups. For the CSQ-8 version, scores range from 8 to 32, with higher values indicating higher satisfaction. Scoring for other versions is similar after extrapolating for number of items.

The following endpoint will be analyzed with CSQ-8 PROMs Questionnaire data.

**Endpoint:** Mean difference in total score using the validated CSQ-8 (Client Satisfaction Questionnaire) administered after treatment at day 90. **Summary measure:** Mean difference in total scores between treatment groups.

#### 2.6.1.2 The PAM PROMs Questionnaire

This study will use the 13-point PAM questionnaire, which will be complimented by data on medication adherence to Inclisiran or standard of care recorded during the trial. The 13 item PAM consists of 13 statements relating to patients beliefs about health care, confidence in their management of health related tasks, and self-assessed knowledge of their condition.

For each statement patients are required to say how much they either agree or disagree on a response scale of 1–4, where 1 represents "strongly disagree" and 4 represents "strongly agree". Patients may also answer "non-applicable" which is scored as 0. A total score is created by summing the scores for the 13 statements and multiplying by 13/(13-n) where n is the number of statements answered as "non-applicable" or missing. The total is rounded to the nearest integer. The total score in the range [13,52] is then converted to a score in the range [0,100] using a calibration table. Note that if n>3, the calibrated score defaults to 51.

The continuous PAM scores are then categorized into four levels for descriptive purposes: according to the materials supplied by Insignia, scores less than 47.1 are level 1, scores between

47.1 and 53.2 are level 2, scores between 53.3 and 70.2 are level 3, and scores above 70.2 are level 4.

The following endpoints will be analyzed with PAM PROMs Questionnaire data.

- Endpoint: Mean difference in total score using the validated Patient Activation Measure (PAM) questionnaire administered after treatment at day 90. Summary measure: Difference between treatment groups in mean change in total scores from baseline to Day 90.
- Endpoint: Measures of adherence to cardiovascular disease self-management using the validated Patient Activation Measure (PAM) questionnaire administered after treatment at day 90 and using assessment of medication adherence during the study period. Summary measure: The frequency and percentages of subjects in the four levels of the PAM scores (below) will be summarized. Note that highly activated patients (level 3 and level 4) are more likely to adhere to cardiovascular self-management and thus medication adherence.
  - Level 1: Disengaged and overwhelmed
  - Level 2: Become aware but still struggling
  - Level 3: Taking action
  - Level 4: Maintaining behaviors and pushinng further

#### 2.6.2 Statistical hypothesis, model, and method of analysis

The key secondary variables will be analyzed as follows:

- Mean difference in total score using the validated CSQ-8 (Client Satisfaction Questionnaire) administered after treatment at day 90 between the groups will be analyzed using ANOVA. The test statistics, mean difference, 95% confidence interval and the p-value obtained using the ANOVA will be presented.
- The comparison between inclisiran and inclisiran + behavioural support also will be done and presented as mentioned above. Inclisiran arm will be considered as control for this analysis.
- The descriptive statistics for the total CSQ score will be provided for each treatment group.
- Mean difference in total score using the validated Patient Activation Measure (PAM) questionnaire administered after treatment from baseline today 90 will be analyzed using ANCOVA model. ANCOVA model which assumes unequal variances for treatment group will be used. The model will include the fixed effects of treatment group with baseline total scores as a covariate. The estimate and corresponding 2-sided 95% confidence intervals of mean difference between treatment groups will be calculated. p-value for hypothesis test for mean difference will also be provided. The FAS will be used for this analysis.
- The comparison between inclisiran and inclisiran + behavioural support also will be done and presented as mentioned above. Inclisiran arm will be considered as control for this analysis.

- Measures of adherence to cardiovascular disease self-management using the validated Patient Activation Measure (PAM) questionnaire administered after treatment at day 90 and using assessment of medication adherence during the study period will be summarized by providing the frequency and percentages of subjects in the four levels of the PAM scores (below) by visit and treatment. Note, highly activated patients (level 3 and level 4) are more likely to adhere to cardiovascular self-management and thus medication adherence.
  - Level 1: Disengaged and overwhelmed
  - Level 2: Become aware but still struggling
  - Level 3: Taking action
  - Level 4: Maintaining behaviors and pushinng further
- Also frequeency and percentage of subjects completed each item of PAM questionnaire will be summarized by visit and treatement.

#### 2.6.3 Handling of missing values

No imputation will be applied if the scores are missing at a visit in any the questionnaire. The proportion of missing data will be included in summaries to aid interpretation.

#### 2.7 Safety analyses

For all safety analyses, the safety set will be used.

Safety summaries (tables, figures) will include only treatment emergent adverse events (i.e. adverse events started after the first dose of study treatment or adverse events that were present prior to start of study treatment but increased in severity during the course of the study). Listings will include all data.

Vital signs values that have complete data and time values will be allocated to pre- or post-dose assessment (as per protocol) based on the actual date/time. For values with missing date/time, scheduled visit date and time will be used. This rule will be applied to data from scheduled visits only. If a measurement scheduled as pre-dose is actually performed post-dose, or vice versa, the data will not be used for by visit/time point summary.

#### 2.7.1 Adverse events (AEs)

The number (and percentage) of participants with TEAEs will be summarized by treatment groups and overall in the following ways:

- By treatment, primary system organ class (SOC) and preferred term (PT).
- By treatment, primary system organ class (SOC), PT and maximum severity.
- By treatment, Standardized MeDRA query (SMQ) and PT.

Separate summaries will be provided for study medication related adverse events, death, serious adverse events, other significant adverse events leading to treatment discontinuation.

Unless otherwise specified, SOCs will be sorted alphabetically and, within each SOC, the PTs will be sorted in descending order of frequency in the total column. A participant with multiple

adverse events within the same PT, the AE will be counted only once. A participant with multiple adverse events within a primary system organ class is only counted once towards the total of the primary system organ class. In case of summary by severity or relationship to study drug, summary will be done using the most severe or related occurrence respectively. Listing of all AEs and SAEs will be provided.

**AE reporting for CT.gov and EudraCT**: For the legal requirements of clinicaltrials.gov and EudraCT, two required tables on treatment emergent adverse events which are not serious adverse events, on treatment emergent serious adverse events and SAE suspected to be related to study treatment will be provided by system organ class and preferred term on the safety set population.

If for a same patient, several consecutive AEs (irrespective of study treatment causality, seriousness and severity) occurred with the same SOC and PT:

- a single occurrence will be counted if there is  $\leq 1$  day gap between the end date of the preceding AE and the start date of the consecutive AE
- more than one occurrence will be counted if there is > 1 day gap between the end date of the preceding AE and the start date of the consecutive AE

For occurrence, the presence of at least one SAE / SAE suspected to be related to study treatment / non SAE has to be checked in a block e.g., among AE's in a  $\leq 1$  day gap block, if at least one SAE is occurring, then one occurrence is calculated for that SAE.

The number of deaths resulting from SAEs suspected to be related to study treatment and SAEs irrespective of study treatment relationship will be provided by SOC and PT.

#### 2.7.1.1 Adverse events of special interest / grouping of AEs

Adverse event of special interest (AESI): The number and percentage of participants who reported TEAEs of special interest will be summarized by PT, treatment group. PTs will be sorted in descending order of frequency in the total column. If a participant reported more than one adverse event with the same PT, the AE will be counted only once. If a participant reported more than one AE within the same AESI, the participant will be counted only once at that AESI. Listing of participants with adverse event of special interest will be provided.

The Compound Case Retrieval Strategy (CRS) will be used to determine the MedDRA search criteria to be used to identify events of special interest.

Adverse event of special interest will include the following:

- Hepatotoxicity (Hepatic events)
- New onset or worsening of diabetis mellitus

For search criteria of AE of special interest, refer to Appendix 5.3.

The most recent list of adverse events of special interest at the time of database lock will be used. CRS listing will be provided.

#### 2.7.2 **Deaths**

Please refer section 2.7.1.

#### 2.7.3 Laboratory data

There are no regular laboratory tests required by this protocol. All blood tests will be performed locally by clinical pathology laboratories, in common with usual practice. Methods for sampling, handling and analysis will be the same as usually applied in routine care.

Abnormal laboratory findings, that are detected during the study or are present at baseline and significantly worsen following study drug administration, and are deemed as clinically significant by the investigator will be recorded as AEs if they lead to treatment discontinuation.

#### 2.7.4 Other safety data

#### 2.7.4.1 Vital signs

Absolute values, change from baseline and percentage change from baseline will be summarized for vital sign parameters by visit, time point and treatment group using overall data.

Baseline and change from baseline in height, will be summarized by visit, treatment group using overall data.

All vital signs data will be listed by treatment group, participant, and visit/time and if ranges are available, abnormalities will be flagged.

#### 2.8 Patient-reported outcomes

#### 2.8.1 The CSQ-8 PROMs Questionnaire

The details about Client Satisfaction Questionnaire (CSQ) and the endpoints were mentioned in section 2.6.1.1. For more details on the questionnaire, please refer to the study protocol.

#### 2.8.2 The PAM PROMs Questionnaire

The details about Patient Activation Measure (PAM) Questionnaire and the endpoints were mentioned in section 2.6.1.2. For more details on the questionnaire, please refer to the study protocol.





#### 2.10.1 Other efficacy data

A capillary blood sample will be taken for immediate analysis of the participants lipid profile for assessment of efficacy. This will be performed at screening/baseline visit, day 90 visit and EOS (day 270) visit in the following:



- Non-HDL (calculated)
- LDL-C calculated using Friedwald

Descriptive summaries by treatment group will be presented.

Line-Plot displaying mean and SE of change from baseline will be provided for all parameters using all available visits.

Descriptive summaries by treatment group will be presented.

Listing of all above endpoints for all available visits will be provided.

The threshold analysis on LDL-C data will be performed. Frequency and percentage of patients with secondary prevention who achieved following threshold targets at day 270 will be provided.

- <1.8 mmol/L (<70 mg/dL)
- <1.4 mmol/L (<55 mg/dL)

# 2.10.2



#### 2.11 Interim analysis

There are no interim analyses planned for this study.

#### 3 Sample size calculation

The primary effectiveness endpoint of the study is percent change of LDL-C from baseline. However, the sample size is driven by patient experience (CSQ-8) and patient activation (PAM); two key secondary outcomes in this trial.

The trial has been powered to detect differences equivalent to a Cohen's effect size of 0.3, approximating a 'small-to-medium' effect in conventional terms

A sample size of 300 patients per arm would be able to detect this effect size with 90% power using a one-sided significance level of 0.025 (this includes a 20% allowance for drop-out in this primary care setting).

This sample size could also detect a reduction of at least 10% change of LDL-C from baseline in the inclisiran group compared to the control group (assuming a standard deviation of 30% in the control group and 20% in the inclisiran group based on observed results from previous inclisiran studies).

The total sample size for the study will be 900 participants.

#### 4 Change to protocol specified analyses

•

## 5 Appendix

#### 5.1 Imputation rules

#### 5.1.1 Study drug

Missing/partial start date or end date of treatment will not be imputed.

#### 5.1.2 AE date imputation

#### 5.1.2.1 AE start date imputation

The following table explains the notation used in the logic matrix. Please note that completely missing start dates will not be imputed.

| | Day | Month | Year |
|----------------------------------|----------|-------|------|
| Partial Adverse Event Start Date | Not used | MON | YYYY |
| Treatment Start Date | Not used | TRTM | TRTY |

The following matrix explains the logic behind the imputation.

| | MON MISSING | MON < TRTM | MON = TRTM | MON > TRTM |
|---|---|---|---|---|
| YYYY MISSING | (1) | (1) | (1) | (1) |
| | No convention | No convention | No convention | No convention |
| YYYY < TRTY | ( 2.a ) | (2.b) | (2.b) | (2.b) |
| | Before Treatment<br>Start | Before Treatment<br>Start | Before Treatment<br>Start | Before Treatment<br>Start |
| YYYY = TRTY | ( 4.a ) | (4.b) | (4.c) | (4.c) |
| | Uncertain | Before Treatment<br>Start | Uncertain | After Treatment<br>Start |
| YYYY > TRTY | ( 3.a ) | (3.b) | (3.b) | (3.b) |
| | After Treatment<br>Start | After Treatment<br>Start | After Treatment<br>Start | After Treatment<br>Start |

Before imputing AE start date, find the AE start reference date.

- If the (imputed) AE end date is complete and the (imputed) AE end date < study drug start date then AE start reference date = min(informed consent date, earliest visit date).
- Else AE start reference date = study drug start date

#### Impute AE start date:

- 1. If the AE start date year value is missing, the date uncertainty is too high to impute a rational date. Therefore, if the AE year value is missing, the imputed AE start date is set to NULL.
- 2. If the AE start date year value is less than the treatment start date year value, the AE started before treatment. Therefore:
  - a. If AE month is missing, the imputed AE start date is set to the mid-year point (01JULYYYY).
  - b. Else if AE month is not missing, the imputed AE start date is set to the mid-month point (15MONYYYY).
- 3. If the AE start date year value is greater than the study drug start date year value, the AE started after treatment. Therefore:
  - a. If the AE month is missing, the imputed AE start date is set to the year start point (01JANYYYY).
  - b. Else if the AE month is not missing, the imputed AE start date is set to the later of (month start point (01MONYYYY), AE start reference date + 1 day).

- 4. If the AE start date year value is equal to the study drug start date year value:
  - a. And the AE month is missing the imputed AE start date is set to the AE reference start date + 1 day.
  - b. Else if the AE month is less than the study drug start month, the imputed AE start date is set to the mid-month point (15MONYYYY).
  - c. Else if the AE month is equal to the study drug start date month or greater than the treatment start date month, the imputed AE start date is set to the later of (month start point (01MONYYYY), AE start reference date + 1 day).

If complete (imputed) AE end date is available and the imputed AE start date is greater than the (imputed) AE end date, then imputed AE start date should be set to the (imputed) AE end date.

#### 5.1.2.2 AE end date imputation

For the purpose of date imputation the treatment follow-up period date is defined as the last available visit date.

- 1. If the AE end date month is missing, the imputed end date should be set to the earliest of the (treatment follow up period date, 31DECYYYY, date of death).
- 2. If the AE end date day is missing, the imputed end date should be set to the earliest of the (treatment follow up period date, last day of the month, date of death).
- 3. If AE year is missing or AE is ongoing, the end date will not be imputed.
- 4. If the imputed AE end date is less than the existing AE start date then use AE start date as AE end date.

#### 5.1.3 Concomitant medication date imputation

#### 5.1.3.1 CM start date imputation

The following table explains the notation used in the logic matrix.

| | Day | Month | Year |
|-----------------------|----------|-------|------|
| Partial CM Start Date | Not used | MON | YYYY |
| Treatment Start Date | Not used | TRTM | TRTY |

The following matrix explains the logic behind the imputation.

| | MON MISSING | MON < TRTM | MON = TRTM | MON > TRTM |
|---|---|---|---|---|
| YYYY MISSING | (1) | (1) | (1) | (1) |
| | Uncertain | Uncertain | Uncertain | Uncertain |
| YYYY < TRTY | ( 2.a ) | (2.b) | (2.b) | (2.b) |
| | Before Treatment<br>Start | Before Treatment<br>Start | Before Treatment<br>Start | Before Treatment<br>Start |
| YYYY = TRTY | ( 4.a ) | (4.b) | ( 4.a ) | (4.c) |
| | Uncertain | Before Treatment<br>Start | Uncertain | After Treatment<br>Start |
| YYYY > TRTY | ( 3.a ) | (3.b) | (3.b) | (3.b) |

| <br>MON MISSING | MON < TRTM | MON = TRTM | MON > TRTM |
|-----------------|-----------------|-----------------|-----------------|
| After Treatment | After Treatment | After Treatment | After Treatment |
| Start | Start | Start | Start |

- 1. If the CM start date year value is missing, the imputed CM start date is set to one day prior to treatment start date.
- 2. If the CM start date year value is less than the investigational study treatment start date year value, the CM started before treatment. Therefore:
  - a. If the CM month is missing, the imputed CM start date is set to the mid –year point (01JULYYYY).
  - b. Else if the CM month is not missing, the imputed CM start date is set to the mid-month point (15MONYYYY).
- 3. If the CM start date year value is greater than the investigational study treatment start date year value, the CM started after treatment. Therefore:
  - a. If the CM month is missing, the imputed CM start date is set to the year start point (01JANYYYY).
  - b. Else if the CM month is not missing, the imputed CM start date is set to the month start point (01MONYYYY).
- 4. If the CM start date year value is equal to the investigational study treatment start date year value:
  - a. And the CM month is missing or the CM month is equal to the treatment start date month, then the imputed CM start date is set to one day prior to treatment start date.
  - b. Else if the CM month is less than the treatment start date month, the imputed CM start date is set to the mid-month point (15MONYYYY).
  - c. Else if the CM month is greater than the treatment start date month, the imputed CM start date is set to the month start point (01MONYYYY).

If complete (imputed) CM end date is available and the imputed CM start date is greater than the (imputed) CM end date, then imputed CM start date should be set to the (imputed) CM end date.

#### 5.2 AEs coding/grading

The MedDRA version which will be available at the time of database lock, will be used for the coding purpose of the adverse events.

#### 5.3 Search criteria for AE of special interest

The Adverse events of special interest (AESIs) based on MedDRA terms are defined in the Case Retrieval Strategy (eCRS). To select the corresponding records from SAS dataset ECRS in Novartis computing environment, use

- Compound name (DRGNAM)="KJX839",
- Compound indication (DRGINDC)="Hypercholesterolemia",
- Records with MDRAVER = 25.0

Safety topics flagged in the eCRS using the safety flag (PSURFL =YES) will be filtered and further safety topics mentioned in section 2.7.1.1 will be considered for analyses.

#### 5.4 **Laboratory parameters derivations**

The following table shows the criteria for clinically notable laboratory values. Not all parameters have notable criteria defined:

Table 5-1 Clinical notable criteria for selected laboratory tests

| Test | Notable post-baseline criteria |
|---|---|
| Glucose, fasting | $\geq$ 5.5 to < 7.0 mmol/L |
| _ | $\geq$ 7.0 mmol/L |
| HbA1c | $\geq 5.7 \%$ to $< 6.5 \%$ ( $\geq 39 \text{ mmol/mol to } < 48$ |
| | mmol/mol) |
| | $\geq$ 6.5 % ( $\geq$ 48 mmol/mol) |

Table 5-2 **Notable Liver function test values** 

| Criterion |
|---|
| ALT > 3 x the upper limit of normal range (ULN) |
| ALT > 5 x ULN |
| ALT > 8 x ULN |
| ALT > 10 x ULN |
| ALT > 20 x ULN |
| AST > 3 x ULN |
| AST > 5 x ULN |
| AST > 8 x ULN |
| AST > 10 x ULN |
| AST > 20 x ULN |
| ALT or AST > 3 x ULN |
| ALT or AST > 5 x ULN |
| ALT or AST > 8 x ULN |
| ALT or AST > 10 x ULN |
| ALT or AST > 20 x ULN |
| Total bilirubin > 2 x ULN |
| TBL >2xULN & DBL >ULN |
| TBL >2xULN & DBL >2xULN |
| ALP > 2 x ULN |
| ALT or AST > 3 x ULN and total bilirubin > 2 x ULN |
| ALT or AST > 5 x ULN and total bilirubin > 2 x ULN |
| ALT or AST > 8 x ULN and total bilirubin > 2 x ULN |
| ALT or AST > 10 x ULN and total bilirubin > 2 x ULN |
| ALT or AST > 20 x ULN and total bilirubin > 2 x ULN |
| ALT or AST > 3 x ULN and Total Bilirubin > 2 x ULN and ALP < 2 x ULN (Hy's law) |

ALT = alanine aminotransferase, AST = aspartate aminotransferase, ALP = alkaline phosphatase, DBL = Direct bilirubin

When a criterion contains multiple laboratory parameters, the criterion will only be considered to have been met when all conditions occur within a 3-day window.

The liver function tests are not required as per the assessment schedule of the protocol. This data collected from EMR based on the availability. Whatever data collected will be presented. Normal ranges provided by medical team will be considered for this analysis since reference ranges are not collected in source data.

#### 5.5 Statistical models

#### 5.5.1 Multiple Imputation Wash-out model

A multiple imputation washout model will be utilized for the primary efficacy analysis of the percentage change in LDL-C from baseline to Day 270 endpoint. The washout model can be thought of as a control-based PMM that will be used to explore the possibility of missing data being MNAR for subjects who discontinued the study early. For subjects who discontinued the study early, their missing values will be imputed under the assumption that their outcome would be similar to those in the control group with similar background characteristics. For subjects in the inclisiran groups only missing Day 270 values will be imputed.

For subjects whose LDL-C values are undetectable i.e., both baseline and post-baseline due to device sensitivity for a lipid parameter in inclisiran groups will be considered as missing and imputed under MAR assumption.

For subjects in the control group, their missing values over all visits after early termination as well as undetectable values including both baseline and post-baseline due to device sensitivity for a lipid parameter will be imputed based on the missing at random (MAR) assumption.

Multiple imputation will be used to account for uncertainty in the imputation process and results from the imputed datasets will be combined using Rubin's method. Further details are provided below.

For the control group the following variables will be included in a multiple imputation procedure (SAS PROC MI), this assumes missing data are MAR:

- Baseline value of efficacy measurement (continuous)
- Observed value of efficacy measurement at Day 90 (continuous)
- Observed value of efficacy measurement at Day 270 (continuous)

For the subjects in the inclisiran group who completed the doses and with intermittent missing as well as undetectable data, the following variables will be included in a multiple imputation procedure (SAS PROC MI), this assumes missing data are MAR:

- Baseline value of efficacy measurement (continuous)
- Observed value of efficacy measurement at Day 90 (continuous)
- Observed value of efficacy measurement at Day 270 from the inclisiran group (continuous)

For the subjects in the inclisiran groups and with missing data at Day 270 which does not includes undetectable data, the following variables will be included in a multiple imputation procedure (SAS PROC MI), this assumes missing data are MNAR:

• Baseline value of efficacy measurement (continuous)

#### 5.5.2 Imputation of undetectable data

For each undetectable LDL-C value, a range is determined based on Friedewald's formula. Below table will provide example range calculation when are distributed in different categories.

Table 5-3 Range determination



As a next step, the undetectable LDL-C values are baseline are imputed to create 500 complete sets of baseline LDL-C values. The imputation is performed by fitting a normal distribution to all available baseline LDL-C values including the LDL-C ranges. The imputed values are obtained by sampling from the posterior predictive distribution. As prior distribution for mean and the standard deviation a normal distribution (mean=0, sd=10) and a half-t-distribution (df=3, scale=2.5) are chosen.

To create 500 complete data sets of baseline and post-baseline LDL-C data sets, the following approach is performed for each of the 500 data sets with complete baseline LDL-C data.

- 1. Fit a Bayesian linear mixed model to all available post-baseline LDL-C data including the LDL-C ranges from Day 90 and Day 270.
  - a. The model includes study arm, visit, and baseline LDL-C as well as all interactions as fixed effects.
  - b. The model includes a normally distributed patient-specific random effect and a normally distributed residual error. The variance of the residual error differs by study arm and visit.

- 2. For the missing values or undetectable LDL-C values of patient *i* at visit *j* in study arm *k* that are imputed under the MAR assumption, the imputed value is drawn from the posterior predictive distribution of the outcome (i.e., LDL-C) of patient *i* at visit *j* in study arm *k*.
- 3. For the missing values of patient *i* at visit *j* in the inclisiran arm that are imputed under the jump-to-reference assumption, the imputed value is drawn from the posterior predictive distribution of the outcome (i.e., LDL-C) of patient *i* at visit *j* whereas the components (e.g., fixed effects and random effects) of the posterior predictive distribution that are associated with the inclisiran arm are replaced by the corresponding value from the placebo arm.

The above imputation will be carried out using R software.

Each of the 500 complete data sets is analyzed with an ANCOVA as specified for the primary analysis. The resulting point estimates will be combined using Rubin's method.

#### 5.6 Rule of exclusion criteria of analysis sets

The protocol deviations (PD) and other criteria leading to complete exclusion from analyses sets are provided in below table, which may be updated prospectively and will be finalized before study DBL.

Table 5-4 Protocol deviation criteria leading to exclusion from analysis sets

| Protocol Deviation | | | Excluding from<br>Analysis set | |
|---|---|---|---|---|
| ID | Desctiption | RAN | FAS | SAF |
| INCL01A | No study informed consent prior to performing study assessments | Х | Х | Х |
| INCL01B | No signed informed consent exists at site | Χ | Х | Х |
| INCL02 | Participant's age < 18 years at screening visit | | | |
| INCL03A | Participant not on statin therapy and intolerance not documented | | | |
| INCL03B | Participant is indicated to have partial statin intolerance but not documented | | | |
| INCL04 | Participant's total cholesterol not available at screening visit or is <4mmol/L (160mg/dL) | | | |
| INCL05 | Participant's lipid-lowering therapy at study entry not stable for ≥ 30 days before screening visit | | | |
| EXCL01 | Participant has medical or surgical history that might limit the individual's ability to take study treatments for the duration of the study and/or put the participant at significant risk | | | |
| EXCL02 | Current or planned renal dialysis or transplantation | | | |

| | Protocol Deviation | | cluding f<br>nalysis s | |
|---|---|---|---|---|
| ID | Desctiption | RAN | FAS | SAF |
| EXCL03 | Participant had acute coronary syndrome or stroke less than 4 weeks before the screening visit | | | |
| EXCL05 | Participant is a female of child-bearing potential and NOT agreeing to either abstinence or, if sexually active, to using effective methods of contraception | | | |
| EXCL06A | Participant confirmed to be pregnant or nursing and randomized | | | |
| EXCL06B | Pregnancy test(s) not performed at screening or randomization visit | | | |
| EXCL07 | Treatment with monoclonal antibodies directed towards PCSK9 initiated at any time during the course of the study | | | |
| EXCL08 | Participant has previous exposure to inclisiran or participation in a randomised study of inclisiran | | | |
| EXCL09 | Participants treated with other investigational medicinal products or devices within 30 days or five half lives (whichever is longer) of the screening visit | | | |
| EXCL10 | Participant who plans to move away from the geographical area where the study is being conducted during the study period | | | |
| EXCL11 | The participant has a triglyceride value of greater than or equal to 4.52 | | | |
| COMD01 | Introduction of new lipid lowering therapy (either different statin or new additional therapy) during the study | | | |
| COMD02 | Treatment with monoclonal antibodies directed towards PCSK9 initiated at any time during the course of the study | | | |
| COMD03 | Another investigational treatment initiated at any time during the course of the study | | | |
| OTH01 | Study treatment given and/or assessment(s) performed after withdrawal of ICF | | | |
| OTH02 | Subject resumes study treatment after pregnancy but continues breast feeding | | | |
| OTH03 | Site closed due to GCP reason | | Х | |
| OTH04 | Scheduled visit missed due to COVID-19 | | | |
| OTH05 | Participant discontinues from study due to COVID-19 situation | | | |
| OTH06 | Assessment / procedure at visits changed due to COVID-19 | | | |
| OTH07 | Drug supply method changed due to COVID-19 | | | |

| | Protocol Deviation | | cluding fi | |
|---|---|---|---|---|
| ID | Desctiption | RAN | FAS | SAF |
| OTH08 | The participant has withdrawn from the Behavioural Support calls so these calls are no longer being made | | | |
| OTH09 | Patient received behavioural support calls when they had not been randomised to receive these | | | |
| OTH10 | Patient did not receive behavioural support calls when they had been randomised to receive these | | | |
| OTH11 | Patient visits have occurred out of visit window and/or the visit is very late | | | |
| OTH12 | Other protocol deviation | | | |
| WITH01 | Participant became pregnant during the course of the study but study treatment was not discontinued | | | |
| WITH02 | Participant has been treated with monoclonal antibodies directed towards PCSK9 but study treatment was not discontinued or re-started | | | |
| WITH03 | Participant has received other investigational treatments but study treatment was not discontinued or re-started | | | |
| WITH04 | Participant had a severe and persistent (>14 days despite appropriate treatment) injection site reaction but study treatment was not discontinued | | | |
| WITH05 | Participant had a confirmed anaphylactic reaction but study treatment was not discontinued | | | |
| TRT01 | Participant was given wrong medication number/pack or administered with study drug that was not stored appropriately or dosed with expired medication | | | |
| TRT02 | Participant was not randomized but took study drug | Χ | Χ | |
| TRT03 | Participant received study drug between screening visit and randomization (Day 1) visit by mistake | | | |
| TRT04 | Missed dosing for any reason other than participant safety or withdrawal (and non-COVID-19 related) | | | |
| TRT05 | Participant did not receive study treatment due to COVID-19 | | | |
| TRT06 | Participant discontinues from treatment due to COVID-19 situation | | | |

#### 6 Reference

CKJX839A1GB01 amended protocol v02 dated 12-Sep-2022.

Attkisson, C. C. & Zwick, R. The client satisfaction questionnaire. Psychometric properties and correlations with service utilization and psychotherapy outcome. Eval. Program Plan. 5, 233–237 (1982)

ICH E9(R1) Harmonized Guideline: addendum on estimands and sensitivity analysis in clinical trials to the guideline on statistical principles for clinical trials. Final version on 20 November 2019.

Hibbard J, Gilburt H. Supporting people to manage their health: An introduction to patient activation. 2014. The King's Fund. 25-12-0016. http://

www.kingsfund.org.uk/publications/supporting-people-manage-their-health

Hibbard J, Mahoney E, Stockard J, Tusler M. Development and testing of a short form of the patient activation measure (PAM). Health Serv Res. 2005; 40(6):1918–30.

Hibbard J, Stockard J, Mahoney E, Tusler M. Development of the Patient Activation Measure (PAM): Conceptualizing and measuring activation in patients and consumers. Health Serv Res. 2004;39(4):1005–26.